CLINICAL TRIAL: NCT05979545
Title: EaRly impAct theraPy With Ceftazidime-avibactam Via rapID Diagnostics Versus Standard of Care Antibiotics and Diagnostics in Patients With Bloodstream Infection, Hospital-acquired Pneumonia or Ventilator-associated Pneumonia Due to Pseudomonas Aeruginosa or Carbapenemase Producing Enterobacterales (RAPID)
Brief Title: EaRly impAct theraPy With Ceftazidime-avibactam Via rapID Diagnostics
Acronym: RAPID
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Pfizer (Industry); Biomerieux inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVANCE-ID 22-002; 23-0135 (Other Grant/Funding Number: PFIZER INC); 225457/Z/22/Z (Other Grant/Funding Number: Wellcome Trust); 20535 (Other: BioMerieux)
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Blood Stream Infections; Ventilator Associated Pneumonia; Healthcare Associated Infection; Carbapenem-Resistant Enterobacteriaceae Infection; Hospital-acquired Pneumonia
Keywords: rapid diagnostics; ceftazidime-avibactam; carbapenemase producing Enterobacterales; hospital-acquired; MDR; AMR; ASP; CRE; BCID2; PN Plus
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection; Healthcare-Associated Pneumonia | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Intervention Model Description: The primary aim is to quantify the combined effect of a PCR-based rapid microbiology diagnostic system and locally adapted antibiotic stewardship on patients with infections due to Pseudomonas aeruginosa or carbapenemase producing Enterobacterales. The combined effect of diagnostics and appropriate antibiotic is the primary focus in the RAPID trial as they are closely interlinked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Samples from patients randomised to the intervention arm will undergo the BioFire FilmArray systems. Patients will be then administered with the study drug, ceftazidime-avibactam when Pseudomonas aeruginosa or carbapenemase producing Enterobacterales detected.
  Interventions: Diagnostic Test: Rapid Diagnostics
- Control (No Intervention): Patients randomised to the control arm, will have samples analysed by clinical microbiology laboratories using standard of care diagnostics. Antibiotics treatment will be administered as per usual institutional practice from hospital supplies.

INTERVENTIONS:
Diagnostic Test: Rapid Diagnostics — Patients randomised to the intervention arm, will have the BioFire Blood Culture Identification 2 Panel (BCID2) used for positive blood cultures and/or the BioFire FilmArray Pneumonia plus PanelPneumonia Panel or Pneumonia plus Panel for respiratory tract specimens if having hospital-acquired pneumonia or ventilator-associated pneumonia. Standard of care diagnostics will also be used. Antibiotic guidelines will be provided to clinicians to aid interpretation of test results and treatment prescription. Ceftazidime-avibactam will be available for targeted use in patients with Pseudomonas aeruginosa or carbapenemase producing Enterobacterales.
  Other Names: BioFire FilmArray BCID2; BioFire FilmArray Pneumonia Plus Panel; BioFire FilmArray Pneumonia Panel
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to propose a seamless intervention linking rapid bacterial isolate identification and antibiotic resistance gene detection and targeted antibiotic prescription to minimise time between infection onset and appropriate treatment in patients with Pseudomonas aeruginosa or carbapenemase producing Enterobacterales infections. This is an investigator initiated trial.

The primary hypothesis is that these interventions will lead to improved clinical outcomes amongst patients with hospital-acquired bloodstream infection, hospital-acquired pneumonia or ventilator-associated pneumonia due to carbapenem non-susceptible Pseudomonas aeruginosa or Enterobacterales, compared to standard antibiotic susceptibility testing.

Patients will be randomised to either a control or intervention arm. Patients randomised to the intervention arm will have relevant specimens analysed by rapid microbiological diagnostics and will have early availability of ceftazidime-avibactam if appropriate. Patients randomised to the control arm, will have samples analysed by clinical microbiology laboratories using standard of care diagnostics. Antibiotics will be available to these patients as per usual institutional practice.

DETAILED DESCRIPTION:
This is an open-label, multinational, randomised, superiority trial. Patients will be randomised to control and intervention arms.

Patients randomised to the intervention arm, will have the BioFire Blood Culture Identification 2 Panel (BCID2) used for positive blood cultures and/or the BioFire FilmArray Pneumonia or Pneumonia plus Panel for respiratory tract specimens if having hospital-acquired pneumonia or ventilator-associated pneumonia. Standard of care diagnostics will also be used. Antibiotic guidelines will be provided to clinicians to aid interpretation of test results and treatment prescription. Ceftazidime-avibactam will be available for targeted use in patients with Pseudomonas aeruginosa or carbapenemase producing Enterobacterales.

Patients randomised to the control arm, will have samples analysed by clinical microbiology laboratories using standard of care diagnostics. Antibiotics will be available to these patients as per usual institutional practice.

The main population that will be recruited in the study will be hospitalised patients with bloodstream infections, hospital-acquired pneumonia or ventilator-associated pneumonia due to Pseudomonas aeruginosa or carbapenemase producing Enterobacterales treated with ceftazidime-avibactam, while the secondary population recruited will be those with multidrug resistant (MDR) Gram-negative bacilli. The enrolment criteria are based on the US Centers for Disease Control and Prevention criteria for healthcare-associated infection surveillance.

Clinical and mortality outcomes will be assessed for 60 days post infection. The infection causing bacterial isolates will be collected for genotypic description via whole genome sequencing. The total target sample size is 1900 participants in the main population over 20 study sites.

ELIGIBILITY:
Inclusion Criteria:

1. patient developed clinical symptoms compatible with bloodstream infection, hospital-acquired or ventilator-associated pneumonia (hospital-acquired and ventilator-associated pneumonia should fulfil US CDC NHSN criteria) AND,
2. an appropriate specimen has been received by the participating laboratory - that is, a blood culture bottle showing Gram negative bacilli or a respiratory sample collected for clinical purposes showing Gram negative bacilli on Gram stain;

Exclusion Criteria:

1. Refractory shock or comorbid condition such that patient not expected to survive more than 48 hours; OR,
2. where the bloodstream infection is thought to be related to a vascular catheter and the catheter is unable to be removed; OR,
3. treatment is not with the intent to cure the infection; OR,
4. patient is incarcerated in a correctional facility; OR,
5. patients previously randomised in this trial within the last 60 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause mortality and/or no improvement in SOFA score at Day 14 post index culture | 14 days post index culture
  Patient has died within 14 days from collection of index microbiology culture from any cause or SOFA score has not improved at Day 14 compared with baseline score on day of collection of index microbiology culture

SECONDARY OUTCOMES:
Clinical response | Day 7 and Day 14 post index culture
  Clinical response at Day 7 and Day 14 post index culture, as determined retrospectively by an adjudication committee
All-cause mortality | Day 14, Day 28, and Day 60 post index culture
  All-cause mortality at Day 14, Day 28, and Day 60 post index culture
Functional outcome | Day 14, Day 28 and Day 60 from collection of index culture
  Functional outcome at Day 14, Day 28 and Day 60 from collection of index culture
Composite outcome | Day 28 from index microbiology culture sample
  Composite outcome measure defined by Desirability of Outcome Ranking (DOOR) at Day 28 from index culture sample
Implementation cost-Health Economics | 60 days since enrolment
  Hospital and ICU level length of stay in the 60 days from randomisation

OTHER OUTCOMES:
Genomics studies | Day 0
  Genotype of the infection causing bacterial isolate, as available through whole genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, Professor, Principal Investigator — National University of Singapore
Locations (4):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung, Xitun District
  - Kaohsiung Medical University Hospital, Kaohsiung City
- Sunpasitthiprasong Hospital, Ubon Ratchathani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided